CLINICAL TRIAL: NCT04912128
Title: Stereotactic Radiosurgery Combination With Anlotinib for Limited Brain Metastases in Non-small Cell Lung Cancer
Brief Title: Stereotactic Radiosurgery Combination With Anlotinib for Limited Brain Metastases in NSCLC
Acronym: AnloSBRT
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Huashan Hospital (Other); Tianjin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AnloSBRT
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Stereotactic Body Radiation Therapy
MeSH Terms: interventions — anlotinib; Angiogenesis Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anlotinib group: Patients in Anlotinib group took Anlotinib 1 week before the MRI-based simulation，12mg/d QD，day1~14, 21d/cycle. All patients received SBRT for brain metastases.
  Interventions: Drug: Anlotinib
- SBRT group: Patients in SBRT group took no anti-angiogenic drugs. All patients received SBRT for brain metastases.

INTERVENTIONS:
Drug: Anlotinib — Anlotinib is a novel multi-target tyrosine Kinase inhibitor that inhibits VEGFR2/3, FGFR1-4, PDGFD α/β, c-Kit and Ret.
  Stereotactic Radiosurgery Stereotactic Radiosurgery as the initial treatment of non small cell lung cancer patients with limited brain metastases
  Other Names: Antiangiogenic agents
  Groups: Anlotinib group

SUMMARY:
The purpose of this study is to determine whether stereotactic radiosurgery combination with Anlotinib could improve the efficacy and outcomes for non-small cell lung cancer with limited brain metastases.

DETAILED DESCRIPTION:
This is a retrospective study. The purpose of this study is to determine whether stereotactic radiosurgery combination with Anlotinib could improve the efficacy and outcomes for non-small cell lung cancer with limited brain metastases. Patients in Anlotinib group took Anlotinib 1 week before the MRI-based simulation，12mg/d QD，day1~14, 21d/cycle. Patients in SBRT group took no anti-angiogenic drugs. All patients received SBRT for brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed as non-small cell lung cancer, with brain metastases and measurable lesions;
2. Patients aged between 18 -80 years; with expected survival time>3 months.
3. Patients with no more than 5 brain metastases
4. Patients with normal organ function within 7 days prior to treatment, the following criteria are met:

   1. blood routine examination criteria : i) hemoglobin (HB) ≥90g/L; ii) absolute neutrophil count (ANC) ≥1.5×10e9/L; iii) platelet (PLT) ≥80×10e9/L; b) biochemical tests meet the following criteria: i) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN, if liver metastasis occurred, ALT and AST ≤5 ULN; iii) serum creatinine (Cr) ≤1.5 ULN or creatinine clearance (CCr) ≥60mL/min;

Exclusion Criteria:

1. Patients who had previously used antiangiogenic agents within 1 month;
2. Patients with small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer);
3. Patient with lung squamous cell carcinoma that involved pulmonary hilar, or non-small cell lung cancer with hemoptysis;
4. Patients with cerebral infarction and cerebral hemorrhage;
5. Patients without perilesional edema；
6. Patients with more than grade 2 (NCI-CTCAE v4.0) acute toxicity reaction due to any previous treatment.
7. Patients with factors that affect oral medication (such as cannot swallow, chronic diarrhea and intestinal obstruction, etc.);
8. Patients with visceral dissemination or severe symptoms, which could cause death in short term;
9. Patients with any other severe and/or uncontrolled disease;
10. Patients who received a surgery, a biopsy or a significant traumatic injury within 1 month;
11. Patients with any signs or medical history of bleeding, unhealed wounds, ulcers or fractures, regardless of the severity;
12. Patients underwent artery or venous thrombotic events within 2 months, such as deep vein thrombosis and pulmonary embolism;
13. Patients with a history of psychotropic medicine abuse and cannot quit or have mental disorders;
14. Patients with disease which will severely endanger their security and could not complete this study, according to the judgement of researchers；

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NSCLC patients with limited brain metastases who received stereotactic radiosurgery with or without Anlotinib treatment.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
PFS | 1 years
  progression-free survival

SECONDARY OUTCOMES:
OS | 1 years
  overall survival
ORR | 3 months
  objective response rate
DCR | 3 months
  disease control rate
iORR | 3 months
  intracranial objective response rate
iPFS | 3 months
  intracranial progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology Cancer Center, Peking University Third Hospital 49# North Garden Rd.,Haidian Dist., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No